CLINICAL TRIAL: NCT02789592
Title: A Randomized Double-Blind, Double-Dummy, Crossover Study to Evaluate the Efficacy and Safety of Prolonged-Release Melatonin and Clonazepam in Patients With Rapid Eye Movement (REM) Sleep Behavior Disorder in Parkinson Disease
Brief Title: Efficacy and Safety of Melatonin PR and Clonazepam in Patients With REM Sleep Behavior Disorder in Parkinson Disease
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Seoul National University Hospital (Other)
Collaborators: Kuhnil Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Principal Investigator, BS Jeon, Professor, Seoul National University Hospital
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: H-1604-134-757
Record Dates: First submitted 2016-05-31; First posted 2016-06-03 (Estimated); Last update posted 2016-06-03 (Estimated); Status verified 2016-06

CONDITIONS: REM Sleep Behavior Disorder; Parkinson Disease
Keywords: REM Sleep Behavior Disorder; Parkinson Disease; Randomized Controlled Trial; Clinical Trial; Melatonin; Clonazepam
MeSH Terms: conditions — REM Sleep Behavior Disorder; Parkinson Disease | interventions — Melatonin; Clonazepam

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (6):
- Group 1 (Experimental): Phase 1: Melatonin PR 2 mg 1 tablet+Clonazepam placebo 1 tablet, 1/day before sleeping for 4 weeks Phase 2: Clonazepam 0.5 mg 1 tablet+Melatonin PR placebo 1 tablet, 1/day before sleeping for 4 weeks Phase 3: Melatonin PR placebo 1 tablet+Clonazepam placebo 1 tablet, 1/day before sleeping for 4 weeks
  Interventions: Drug: Melatonin PR; Drug: Clonazepam; Drug: Melatonin PR placebo; Drug: Clonazepam placebo
- Group 2 (Experimental): Phase 1: Clonazepam 0.5 mg 1 tablet+Melatonin PR placebo 1 tablet, 1/day before sleeping for 4 weeks Phase 2: Melatonin PR placebo 1 tablet+Clonazepam placebo 1 tablet, 1/day before sleeping for 4 weeks Phase 3: Melatonin PR 2 mg 1 tablet+Clonazepam placebo 1 tablet, 1/day before sleeping for 4 weeks
  Interventions: Drug: Melatonin PR; Drug: Clonazepam; Drug: Melatonin PR placebo; Drug: Clonazepam placebo
- Group 3 (Experimental): Phase 1: Melatonin PR placebo 1 tablet+Clonazepam placebo 1 tablet, 1/day before sleeping for 4 weeks Phase 2: Melatonin PR 2 mg 1 tablet+Clonazepam placebo 1 tablet, 1/day before sleeping for 4 weeks Phase 3: Clonazepam 0.5 mg 1 tablet+Melatonin PR placebo 1 tablet, 1/day before sleeping for 4 weeks
  Interventions: Drug: Melatonin PR; Drug: Clonazepam; Drug: Melatonin PR placebo; Drug: Clonazepam placebo
- Group 4 (Experimental): Phase 1: Melatonin PR 2 mg 1 tablet+Clonazepam placebo 1 tablet, 1/day before sleeping for 4 weeks Phase 2: Melatonin PR placebo 1 tablet+Clonazepam placebo 1 tablet, 1/day before sleeping for 4 weeks Phase 3: Clonazepam 0.5 mg 1 tablet+Melatonin PR placebo 1 tablet, 1/day before sleeping for 4 weeks
  Interventions: Drug: Melatonin PR; Drug: Clonazepam; Drug: Melatonin PR placebo; Drug: Clonazepam placebo
- Group 5 (Experimental): Phase 1: Clonazepam 0.5 mg 1 tablet+Melatonin PR placebo 1 tablet, 1/day before sleeping for 4 weeks Phase 2: Melatonin PR 2 mg 1 tablet+Clonazepam placebo 1 tablet, 1/day before sleeping for 4 weeks Phase 3: Melatonin PR placebo 1 tablet+Clonazepam placebo 1 tablet, 1/day before sleeping for 4 weeks
  Interventions: Drug: Melatonin PR; Drug: Clonazepam; Drug: Melatonin PR placebo; Drug: Clonazepam placebo
- Group 6 (Experimental): Phase 1: Melatonin PR placebo 1 tablet+Clonazepam placebo 1 tablet, 1/day before sleeping for 4 weeks Phase 2: Clonazepam 0.5 mg 1 tablet+Melatonin PR placebo 1 tablet, 1/day before sleeping for 4 weeks Phase 3: Melatonin PR 2 mg 1 tablet+Clonazepam placebo 1 tablet, 1/day before sleeping for 4 weeks
  Interventions: Drug: Melatonin PR; Drug: Clonazepam; Drug: Melatonin PR placebo; Drug: Clonazepam placebo

INTERVENTIONS:
Drug: Melatonin PR — For experimental treatment of RBD
  Other Names: Circadin
Drug: Clonazepam — For experimental treatment of RBD
  Other Names: Rivotril
Drug: Melatonin PR placebo — Placebo pill manufactured to mask melatonin PR 2mg tablet
  Other Names: Placebo tablet of Melatonin PR
Drug: Clonazepam placebo — Placebo pill manufactured to mask clonazepam 0.5mg tablet
  Other Names: Placebo tablet of clonazepam

SUMMARY:
The purpose of this study is to determine whether melatonin prolonged-release (PR) and clonazepam are effective and safe in the treatment of rapid eye movement behavior disorder (RBD) of patients with Parkinson's disease (PD).

DETAILED DESCRIPTION:
RBD is one of the representative non-motor symptoms of PD. Patients with RBD show dream-enacting behaviors such as punching, kicking, singing, screaming, or somnambulism. These can interfere in sleep quality and increase the risk of falling down from the bed and physical injuries of both the patient and sleep partner. Therefore, qualities of life of the patient and sleep partner are negatively influenced by presence of RBD.

Clonazepam has been used for treatment of choice of RBD. However, the efficacy of clonazepam is not proven in the clinical trial. Clonazepam has several side effects that could be problematic in PD patients such as increasing fall-down risk, daytime somnolence, and cognitive decline. Melatonin is a second-line treatment option for RBD, but there has been only one randomized crossover trial that evaluated the efficacy of melatonin on RBD. Finally, there has been no study that evaluate and compare the efficacy and safety of melatonin and clonazepam for treatment of RBD.

ELIGIBILITY:
Inclusion Criteria:

* Subject was enrolled voluntarily and understood the contents of this clinical trial
* Subject was diagnosed as Parkinson disease (PD)
* Hoehn and Yahr (H&Y) stage 1, 2, or 3
* Existence of caregivers who can provide a information about symptoms of rapid eye movement sleep disorder (RBD) of the participant
* RBD frequency is one or more per week
* Existence of RBD by answering "yes" to the question (RBD-1Q): "Have you ever been told, or suspected yourself, that you seem to 'act out your dreams' while asleep (for example, punching, flailing your arms in the air, making running movements, etc.)?"
* Good compliance for reporting PGI scores and sleep diary

Exclusion Criteria:

* Existence of cognitive decline hard to participate in the clinical trial
* Hypersensitivity to melatonin or clonazepam
* Previous melatonin or clonazepam treatment within 1 month
* Changing anti-parkinsonian medications within 1 month
* Current treatment with sedatives or hypnotics at bedtime
* Diagnosed as epilepsy or current treatment with anti-epileptic drugs
* Severe trauma history due to RBD
* Lactating, pregnant, or possible pregnant
* Subject has confusion or visual hallucination in daytime
* Diagnosed as obstructive sleep apnea or severe snoring
* Diagnosed as other parasomnia
* Presence of severe psychiatric illness
* Alcoholics or drug abuser
* Myasthenia gravis
* Acute narrow-angle glaucoma
* Prior participation to other clinical trials within 3 months
* Presence of severe comorbidities or a cancer
* Existence of illness or problems which makes difficult to be enrolled to this trial judged by clinicians

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2016-07; Primary Completion 2019-12 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Clinical Global Impression-Improvement scale (CGI-I) | Four weeks (plus or minus 3 days)
  Clinician assessed rating scale of clinical improvement or worsening relative to a baseline state, scored as 1, very much improved; 2, much improved; 3, minimally improved; 4, no change; 5, minimally worse; 6, much worse; or 7, very much worse.

SECONDARY OUTCOMES:
Mean change of the Clinical Global Impression-Severity scale (CGI-S) | Four weeks (plus or minus 3 days)
Patient Global Impression-Improvement scale (PGI-I) | Four weeks (plus or minus 3 days)
Mean change of the Patient Global Impression-Severity scale (PGI-S) | Four weeks (plus or minus 3 days)
modified RBD Questionnaire-HongKong (mRBDQ-HK) | Four weeks (plus or minus 3 days)
Mean change of the Epworth Sleepiness Scale (ESS) | Four weeks (plus or minus 3 days)
Mean change of the Parkinson Disease Sleep Scale (PDSS) | Four weeks (plus or minus 3 days)
Mean change of the Montreal Cognitive Assessment (MoCA) | Four weeks (plus or minus 3 days)
Mean change of the Unified Parkinson's Disease Rating Scale (UPDRS) | Four weeks (plus or minus 3 days)
Sleep diary | Four weeks (plus or minus 3 days)

CONTACTS AND LOCATIONS:
Overall Officials: Beomseok Jeon, MD, PhD, Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Arnulf I. REM sleep behavior disorder: motor manifestations and pathophysiology. Mov Disord. 2012 May;27(6):677-89. doi: 10.1002/mds.24957. Epub 2012 Mar 22. PMID 22447623
- [Background] Sixel-Doring F, Trautmann E, Mollenhauer B, Trenkwalder C. Associated factors for REM sleep behavior disorder in Parkinson disease. Neurology. 2011 Sep 13;77(11):1048-54. doi: 10.1212/WNL.0b013e31822e560e. Epub 2011 Aug 10. PMID 21832215
- [Background] Kunz D, Mahlberg R. A two-part, double-blind, placebo-controlled trial of exogenous melatonin in REM sleep behaviour disorder. J Sleep Res. 2010 Dec;19(4):591-6. doi: 10.1111/j.1365-2869.2010.00848.x. PMID 20561180
- [Background] Schenck CH, Montplaisir JY, Frauscher B, Hogl B, Gagnon JF, Postuma R, Sonka K, Jennum P, Partinen M, Arnulf I, Cochen de Cock V, Dauvilliers Y, Luppi PH, Heidbreder A, Mayer G, Sixel-Doring F, Trenkwalder C, Unger M, Young P, Wing YK, Ferini-Strambi L, Ferri R, Plazzi G, Zucconi M, Inoue Y, Iranzo A, Santamaria J, Bassetti C, Moller JC, Boeve BF, Lai YY, Pavlova M, Saper C, Schmidt P, Siegel JM, Singer C, St Louis E, Videnovic A, Oertel W. Rapid eye movement sleep behavior disorder: devising controlled active treatment studies for symptomatic and neuroprotective therapy--a consensus statement from the International Rapid Eye Movement Sleep Behavior Disorder Study Group. Sleep Med. 2013 Aug;14(8):795-806. doi: 10.1016/j.sleep.2013.02.016. Epub 2013 Jul 22. PMID 23886593